CLINICAL TRIAL: NCT00242164
Title: Defining The Role Of Dialysate Magnesium In Arrhythmogenicity On Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Renal Research Institute (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DRDA 05-2076
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2005-07

CONDITIONS: Chronic Kidney Disease; Arrhythmia
Keywords: Hemodialysis; Magnesium; Arrhythmia; QTc interval; QT dispersion
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arrhythmias, Cardiac

INTERVENTIONS:
Drug: Dialysate Magnesium (Concentration)

SUMMARY:
The study is being performed to better understand dialysis techniques which keep heart functions stable during dialysis. People on dialysis have a high risk for heart disease and strokes. More information about dialysis techniques that keep hearts stable may help prevent the high risk of cardiovascular disease and death and help to reduce discomfort during dialysis. This study will look at the way that the magnesium in dialysate affects heart function during dialysis. High or low levels of magnesium may change the way hearts beat. The question asked is if lowering the amount of magnesium in dialysate will affect the amount of magnesium in blood or change the heart beat.

DETAILED DESCRIPTION:
Heart disease is a major cause of illness and death among patients on dialysis. Changes in the heart's rhythm and sudden cardiac death are also important problems in this group. Abnormal rhythm can occur during hemodialysis.

During dialysis, the blood comes in contact with a solution called dialysate. This solution contains minerals like calcium, potassium and magnesium. Some studies have indirectly suggested that lower magnesium in dialysis patients protects them from having rhythm problems.

Factors that increase the chance for the development of abnormal rhythms can be indirectly assessed by evaluating the electrocardiogram (EKG). This is done by measuring the distance between the wave forms on the EKG. One of these is called the QT interval. QT dispersion is a value derived from the QT interval. A long QT interval is thought to make an individual more prone to having abnormal heart rhythms.

Therefore it is planned to study the effect of low levels of magnesium in the dialysate on QT interval and dispersion and the tendency for rhythm change. QT interval changes will be compared during dialysis with low magnesium with QT interval changes during dialysis with normal magnesium.

This will be a cross over trial including 24 adult male and female patients on chronic hemodialysis. Subjects will be studied during two of their regular dialysis sessions, the only difference being the amount of magnesium in the dialysate. QT interval and QT dispersion will be calculated from the EKG recordings before and after each dialysis session.

The results of this study will lead to a better understanding of cardiovascular risks in patients undergoing chronic dialysis and may offer a potentially novel strategy to reduce the risk of abnormal heart rhythms risk during dialysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over with end-stage renal disease. (ESRD)
* have been on maintenance hemodialysis therapy three times/week for greater than or equal to 3 months
* All causes of renal failure are included

Exclusion Criteria:

* less than 18 years of age
* have been on maintenance hemodialysis therapy three times/week for less than 3 months
* are pregnant or lactating
* unable or unwilling to provide informed consent
* currently participating in a clinical trial with an intervention
* systolic (top number) blood pressure levels greater than or equal to 180 or less then 80
* diastolic (bottom number) blood pressure levels greater than 110
* a hemoglobin level (red blood cell measure) that is less than 8mg/dl
* a corrected calcium level that is greater than 11mg/dl or less than 8mg/dl
* had a change in their anti-hypertensive medications within the last three weeks
* clinical signs and symptoms of untreated or unresolved infection
* clinical evidence requiring admission to the hospital
* had a cerebral vascular accident or myocardial incident within the past 3 months
* Based on the assessment of the investigators, or study coordinator designee, patients who appear unlikely or unable to participate in the required study procedures
* Patients with a history of arrhythmias, recent electrophysiological evaluation and or having pacemakers are excluded.
* Patients with acute renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2005-11; Primary Completion 2006-06 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the difference in QT dispersion between low dialysate magnesium and normal dialysate magnesium | over one dialysis session
  measurement will be the duration of some changes in the EKG.

CONTACTS AND LOCATIONS:
Overall Officials: Panduranga S Rao, MD, DNB, MS, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan Dialysis Center, Ann Arbor, Michigan
  - University of Michigan Dialysis Center, Livonia, Michigan

REFERENCES:
- See also: Dr. Panduranga Rao's University of Michigan webpage — http://www.med.umich.edu/intmed/nephrology/STAFF/rao_ps1.htm